CLINICAL TRIAL: NCT02876198
Title: Study of the Modification of the Retinal Nerve Fiber Layer in Patients Treated With Intravitreous Injection of Anti-VEGF
Acronym: IVT-RNFL
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2015_41
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Retinal Neovascularization
Keywords: Retinal neovascularization; Anti-VEGF; Retinal Nerve Fiber Layer (RNFL)
MeSH Terms: conditions — Retinal Neovascularization | interventions — Gonioscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients treated with anti-VEGF
  Interventions: Device: Gonioscopy

INTERVENTIONS:
Device: Gonioscopy — Study of the trabecular structure by gonioscopy

SUMMARY:
The intra-vitreous injection (IVT) of anti-VEGF (vascular endothelial growth factor) is currently the standard treatment for retinal neovascularization. The VEGF stimulates endothelial cells' proliferation and migration. It also increases microvascular permeability. If the VEGFs have proven their efficiency in the decrease of choroidal neovascular proliferation, their impact of the head of the optic nerve's microvasculature is yet unknown. Knowing that this microvasculature provides the retinal nerve fibers with oxygen, located in the area of the head of the optic nerve, a vasoconstriction induced by the anti-VEGF may have an incidence on the loss of retinal nerve fibers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patients treated with anti-VEGF according to the French summary of product characteristics (SPC)
* Patients who have been informed of the trial and who are not opposed to participate in the study

Exclusion Criteria:

* Patients presenting a retinal condition, including the optic nerve
* Patients treated with anti-VEGF in both eyes
* Pregnant women
* Lack of affiliation to social security or universal health coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during a consultation in ophtalmology after prescription of an anti-VEGF treatment.
  The study will not change the patient's usual care schedule. Only a different analysis of the images obtained by SD -OCT will be performed, and a gonioscopy will be carried out systematically the inclusion of patient and 12 months.
  The data for the study will be collected at the inclusion visit and at the final visit of the study at 12 months.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
change in RNFL's thickness in the nasal quadrant of the optic nerve after intra-vitreous Injection of Anti-VEGF | Change from baseline RNFL's thickness at Month 12
  RNFL's thickness (in microns) measured with the Heildelberg glaucoma module of the spectral domain Optical Cohérence Tomographie (OCT Spectralis, Heidelberg engeening).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Pole Vision du val d'Ouest, Lyon
  - Fondation Ophtalmologique A. de Rotchschild, Paris
  - Centre médical et chirurgical de la rétine, Strasbourg